CLINICAL TRIAL: NCT06548594
Title: Out-of-State, At-Home, Transcutaneous Auricular Neuromodulation for Hypermobile Ehlers Danlos Syndrome
Brief Title: Out of State - tAN hEDS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: MUSC Blue Sky initiative (Unknown)
Responsible Party: Principal Investigator, Jeffrey Borckardt, Associate Professor-Faculty, Medical University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00138254
Record Dates: First submitted 2024-08-07; First posted 2024-08-12 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-10

CONDITIONS: Hypermobile EDS (hEDS)
Keywords: Brain
MeSH Terms: conditions — Ehlers-Danlos syndrome type 3

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Four Weeks of Active Transcutaneous Auricular Neurostimulation (Experimental): Participants will receive 4 weeks of at-home, self-administered active Transcutaneous Auricular Neurostimulation (tAN).
  Interventions: Device: Transcutaneous Auricular Neurostimulation

INTERVENTIONS:
Device: Transcutaneous Auricular Neurostimulation — Transcutaneous Auricular Neurostimulation (tAN) is a wearable, electrical stimulation device that delivers electricity to specific parts of the human ear.

SUMMARY:
Hypermobile EDS and hypermobile spectrum disorder (collectively referred to as hEDS) are estimated to affect 1 in 500 individuals worldwide. hEDS patients have limited treatment options for their numerous symptoms that impact the quality of life. This clinical trial tests a new ear stimulation method in hEDS patients to determine if it may improve quality of life.

DETAILED DESCRIPTION:
The Ehlers-Danlos syndromes (EDS) are a group of heritable, connective tissue disorders characterized by joint hypermobility, skin hyperextensibility, and tissue fragility2. Hypermobile EDS (hEDS) is the most common type of EDS and is estimated to affect 1 in 500 individuals worldwide1. Note that there are specific clinical criteria for hEDS and those who do not meet all of them but have a number of similar symptoms are usually classified with hypermobility spectrum disorder (HSD). When investigators use the term hEDS investigators include those with HSD as well. hEDS is characterized by broad tissue/organ involvement across multiple systems and incomplete penetrance. Of particular interest for the proposed work, the vagus nerve has afferent and efferent interactions with nearly all of the affected systems (i.e., cardiovascular, GI, immune system, neurologic function). hEDS is a chronic and debilitating disease that oftentimes begins during childhood and worsens at the time of puberty3. In general, hEDS affects women more severely than men and they are more frequently diagnosed. Treatment options are limited to symptom management and may include physical therapy, bracing and mobility aids, pain management and medication for co-morbid conditions. Surgical intervention is frequent in hEDS patients with an average of 4-5 surgeries required prior to the age of 25 and some are left bed bound and severely handicapped. According to recent reports, 50% of hEDS patients have considered suicide due to not only chronic pain, depression and surgeries, but sadly due to physician-patient interactions being dismissive.

hEDS is viewed as the most neglected disease in modern medicine. The healthcare burden is significant with annual costs estimated at ~$100K/year/patient with a total cost of $3-10M over a lifetime per patient. Physicians are taught limited and misleading information in medical school that Ehlers Danlos Syndromes are benign and rare diseases. These education deficiencies combined with phenotype heterogeneity result in diagnostic challenges. Consequentially, the average time to diagnosis from first symptoms is 14 years. The proposed studies in this application are an important step in transforming how the disease is viewed and understood in the medical community and will provide hope to the many patients with hEDS.

As there is little known about the etiology of the multi-system dysfunction and co-morbidities in hEDS, investigators propose an exploratory study of wide breadth to search for the most promising follow-up investigations. To that end, our main goal is to establish a human trial to investigate the effect of hEDS on multiple body systems and the potentially beneficial effects of an intervention known to have effects on most of those same body systems (vagus nerve stimulation - VNS). Investigators propose to advance mechanistic understanding of hEDS and to test a new therapeutic approach.

Specific Aim: Investigate whether 4 weeks of at-home transcutaneous auricular VNS (tAN) improves a battery of nine key physical and psychological symptoms of a group of hEDS patients (n=36) using an open-label active only design. Investigators will remotely collect clinical measures at baseline, and weekly timepoints through week 4, as well as a 3 month follow up. Investigators will test patients in the following domains: pain, fatigue, sleep, anxiety, depression, quality of life, GI function, immune function and autonomic function.

ELIGIBILITY:
Inclusion Criteria:

* Ages of 18 and 65;
* Participants who meet the 2017 diagnostic criteria for hEDS or HSD4-5 with persistent symptoms in at least two of the domains to be followed during the intervention (pain, fatigue, sleep, anxiety, depression, quality of life, GI function, autonomic function and immune function)
* Mentally capable of reading, writing, giving consent, and following instructions;

Exclusion Criteria:

* Mentally capable of reading, writing, giving consent, and following instructions;
* Not pregnant;
* No history of seizures;
* no prior history of trauma or damage to ear
* History of documented Autism spectrum disorder (ASD) diagnosis
* Residing in the state of South Carolina

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-11-27 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Ehlers-Danlos Syndrome Symptom Battery | 4 weeks
  The investigators have created an Ehlers-Danlos Syndrome Symptom Battery that measures a variety of different primary and secondary symptoms associated with Ehlers-Danlos Syndrome, including: Pain, Fatigue, Sleep, Anxiety, Depression, Quality of Life, and Gastrointestinal issues.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Borckardt, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina Institute of Psychiatry, Charleston, South Carolina, United States